CLINICAL TRIAL: NCT01831596
Title: Evaluation of a Novel Post-Surgical Dressing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated by Spiracur. Efforts were made to contact the PI/study team members, but were unsuccessful.
Sponsor: KCI USA, Inc (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030110
Record Dates: First submitted 2013-04-05; First posted 2013-04-15 (Estimated); Results first posted 2020-09-28 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Post Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ciSNaP (Experimental)
  Interventions: Device: ciSNaP

INTERVENTIONS:
Device: ciSNaP — SNaP disposable, mechanically powered Negative Pressure Wound Therapy System

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Closed-Incision SNaP Device.

ELIGIBILITY:
Inclusion Criteria:

* Surgically closed incision.
* Subject is 18 years of age or older.
* Subject consents to follow-up per protocol.
* Willing and able to sign informed consent.

Exclusion Criteria:

* Subject is allergic to wound care products used in this study.
* Subject has wounds with exposed blood vessels not suitable for negative pressure therapy.
* Pregnant or pregnancy-suspected subject.
* Subject actively participating in other clinical trials that conflict with the current study.
* Subject is unable or unwilling to comply with protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- El Camino Hospital, Mountain View, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ciSNaP
Started | 59
Completed | 51
Not Completed | 8
Not completed — Other | 8

BASELINE CHARACTERISTICS:
Arm/Group | ciSNaP
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity (White) | 41
  Ethnicity (Non-White) | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Complaints About Device Use and Operation
Description: Frequency of complaints about device use and operation
Time Frame: 30 days
Population: The study was terminated by Spiracur. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Arm/Group | ciSNaP
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | ciSNaP
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 6/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ciSNaP (N=51)
Blister (Skin and subcutaneous tissue disorders) | 2 (2)
Mild surgical infection (Infections and infestations) | 2 (2)
Congestive Heart Failure exacerbation (Cardiac disorders) | 1 (1)
Stitch granuloma (Skin and subcutaneous tissue disorders) | 3 (3)
Minor dehiscence (Skin and subcutaneous tissue disorders) | 3 (3)
Hemarthrosis (Blood and lymphatic system disorders) | 1 (1)
Lymphocele (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No